CLINICAL TRIAL: NCT05512754
Title: Randomized Controlled Trial of Anti-inflammatory Medications in Patients With Elevated Serum Prostate-specific Antigen
Brief Title: Impact of Anti-inflammatory Medications in Patients With Elevated Serum Prostate-specific Antigen
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-1952
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Elevated Serum PSA
Keywords: PSA
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Randomization into two groups between Group A (No NSAIDs) or Group B (Ibuprofen 400 mg q 8 h for 10 days)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibuprofen (Experimental): Participants receive Ibuprofen 400 mg tablet orally every 8 hours for 10 days
  Interventions: Drug: Ibuprofen 400 mg
- Control (No Intervention): Participants receive no NSAIDs

INTERVENTIONS:
Drug: Ibuprofen 400 mg — 400 mg tablet
  Other Names: Advil
  Arms: Ibuprofen

SUMMARY:
The purpose of this study is to assess the impact of ibuprofen in men with elevated serum PSA.

DETAILED DESCRIPTION:
Serum prostate-specific antigen (PSA) is widely used as a screening marker for prostate cancer. However, elevated serum PSA level could result from various conditions other than malignancy such as benign prostatic hyperplasia (BPH), urinary tract infection, or inflammation (prostatitis). Inflammation within the prostate is often sub-clinical, not readily visible on urinalysis, and can putatively and artificially elevate PSA. Non-steroidal anti-inflammatory drugs (NSAIDs) have shown benefits in reducing symptoms in patients with inflammatory conditions of the prostate. Ibuprofen (Advil, Motrin) is a widely available, cheap, and commonly used over the counter NSAID. NSAID's are routinely given to men with an elevated PSA for empiric treatment of inflammation; however, the impact of NSAIDs in men with elevated serum PSA is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Male patients age between 18-80 years old with a screening PSA > 3 ng/ml being considered for additional diagnostic testing (e.g., MRI, biopsy)
* Normal digital rectal examination.
* No clinical symptoms concerning acute urinary tract infection (e.g. dysuria, malodorous urine, positive urine culture)

Exclusion Criteria:

* Active urinary tract infections or bacteriuria
* Known prostate cancer
* Urethral catheter within the last 6 weeks
* History of hypersensitivity or allergy to ibuprofen or NSAIDs.
* Known severe chronic kidney disease: eGFR < 30 mL/min/1.73 m2
* Known history of severe liver disease (elevated AST or ALT greater than 3 times upper limit of normal)
* History of gastrointestinal bleeding or NSAIDs induced GI adverse events
* Concomitant dual-antiplatelet use or anticoagulants
* Concomitant anti-inflammatory or steroidal drugs
* Known bleeding disorder(s)
* Patients with a solitary kidney or history of a kidney transplant
* Any other medical contraindication to NSAIDs

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of serum PSA compared with baseline | Baseline, 6 weeks
  serum prostatic specific antigen

SECONDARY OUTCOMES:
Change of International Prostate Symptom Score (IPSS) compared with baseline | Baseline, 6 weeks
  Self-reported questionnaires measured lower urinary tract symptoms ranging from 0 to 35.
  Higher score mean worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Eggener, MD, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - Albany Medical College, Albany, New York
  - The Pennsylvania State University at The Milton S. Hershey Medical Center, Hershey, Pennsylvania

REFERENCES:
- [Background] Josefsson A, Mansson M, Kohestani K, Spyratou V, Wallstrom J, Hellstrom M, Lilja H, Vickers A, Carlsson SV, Godtman R, Hugosson J. Performance of 4Kscore as a Reflex Test to Prostate-specific Antigen in the GOTEBORG-2 Prostate Cancer Screening Trial. Eur Urol. 2024 Sep;86(3):223-229. doi: 10.1016/j.eururo.2024.04.037. Epub 2024 May 20. PMID 38772787
- [Background] Aguiar JA, Li EV, Ho A, Bennett R 4th, Li Y, Neill C, Schaeffer EM, Patel HD, Ross AE. Ultrasensitive PSA: rethinking post-surgical management for node positive prostate cancer. Front Oncol. 2024 Apr 9;14:1363009. doi: 10.3389/fonc.2024.1363009. eCollection 2024. PMID 38655143